CLINICAL TRIAL: NCT04280315
Title: Investigation of the Skin Barrier in Patients With Type 1 Diabetes - a Case-control Study
Brief Title: Investigation of the Skin Barrier in Patients With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Jannet Svensson (Other)
Responsible Party: Sponsor-Investigator, Jannet Svensson, MD, PhD, Assistant Professor, Copenhagen University Hospital at Herlev
Organization: Copenhagen University Hospital at Herlev (Other)
Other Study IDs: SkinBarrier_30092019
Record Dates: First submitted 2020-02-14; First posted 2020-02-21 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Type 1 Diabetes
Keywords: Dermatology; Skin Barrier Function
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Buccal Swab for DNA extraction
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Cases are patients with type 1 diabetes in three age strata:
  * 20 participants in the age of 2-10 years
  * 20 participants in the age of 11-20 years
  * 10 participants with more than 30 years of diabetes duration
- Controls: Controls are age and sexmatched with the cases and are recruited from the neuropediatric clinic at Herlev Hospital as well as relatives and parents of patients in the whole Pediatric Department

SUMMARY:
This study is a case-control study comparing the skin barrier between 50 T1D patients with healthy controls in 3 age-strata including both pediatric and adult patients.

DETAILED DESCRIPTION:
The skin is a crucial barrier against external allergens and irritants. Therefore the function of the skin barrier is central regarding evolvement of eczema. In patients with type 1 diabetes (T1D) using insulin pumps and/or glucose sensor, eczema is unfortunately a frequent reaction. The skin consists of three layers: epidermis, dermis and subcutaneous fat, whereas epidermis is most determining regarding skin barrier. Epidermis can further be subdivided, where stratum corneum (SC) is the outer part, which means most regarding vulnerability towards external allergens.

The function of the skin barrier can be investigated by non-invasive methods using transepidermal water loss (TEWL), which shows the water vapour flux from the skin. Besides SC can be determined using the tape strip method, where few SC cells are peeled off and thereby can be analyzed with mass-spectrometry. Natural moisturizing factors (NMF) is though one of the very important functionalities of the SC, which are determined by the amount of 2-pyrrolidone-5-carboxylic acid (PCA). Besides, the lipid distribution, presence of antimicrobial peptide and cytokine response give as well important information regarding the skin barrier.

Dermatological manifestations of T1D are quite frequent and have been shown to be related to glycemic control, placing dermatological manifestations as a precursor of other microvascular complications11. There is a lack of studies regarding skin barrier function in patients with T1D, and especially in a pediatric study population. Therefore, this case-control study will be conducted investigating skin barrier function in pediatric patients with T1D compared to healthy controls in order to both meet this lack of knowledge, but as well to improve the prevention of skin problems to devices used in T1D-treatment.

The examination program of just one visit per participant consists of:

* TEWL-measure at forearm and buttock
* Buccal swab regarding filaggrin gene status
* Microbiological swab from the skin at forearm and buttock
* 2X11 tape strips from the skin at foream and buttock to be analyzed for NMF, Lipid, Cytokines, Antimicrobial peptide and Dermal Topographical Index as well as protein content using SquameScan
* Measure of skin PH, hydration and sebum content at forearm and buttock
* Capillary Blood Glucose
* Survey regarding atopic and dermatological symptoms

ELIGIBILITY:
Cases:

Inclusion Criteria:

* Diagnosed with type 1 diabetes, more than 6 months ago

Exclusion Criteria:

* Skin lesions at both buttocks and forearms so investigation can not be done
* Known skin diseases with decreased barrier function like atopic dermatitis, psoriasis and allergic contact dermatitis
* Active infectious disease
* Use of immunosuppressive medication e.g. steroids
* Lack of language competence in Danish

Controls:

Inclusion Criteria:

* Diagnosed with Tourettes or Headache OR sibling for patients in the 1813-clinic at Pediatric Emergency Toom OR Hospitalized patients at Pediatric department OR Parents to alle these

Exclusion Criteria are equal to exclusion criteria in cases

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study Population are included from the Pediatric department in the diabetes group for patients and primarily in the neurogroup for controls. Adult cases are included from Steno Diabetes Center Copenhagen and adult controls as parents to patients included.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
TEWL | Baseline
  Transepidermal Water Loss measured by an Aquaflux AF1000

SECONDARY OUTCOMES:
Skin barrier properties described with Tape Strips | Baseline
  Tape strips will be analyzed according to Natural Moisturizing Factors
Filaggrin mutation Status | Baseline
  Filaggrin DNA status regarding common SNPs in DNA
Skin pH | Baseline
  Measured with DermaUnit SSC3 Skin pH-Meter
Skin hydration | Baseline
  Measured with DermaUnit SSC3 Corneometer
Sebum content in skin | Baseline
  Measured with DermaUnit SSC3 Sebumeter

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Steno Diabetes Center Copenhagen, Gentofte Municipality, Capital Region
  - Department of Pediatrics, Herlev Hospital, Herlev, Capital Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.herlevhospital.dk/afdelinger-og-klinikker/Afdeling-for-Boern-og-Unge/Forskningsprojekter/Sider/Diabetes/Hudproblemer-i-forbindelse-med-insulinpumpe-og-sensor.aspx